CLINICAL TRIAL: NCT00889304
Title: Study on Quality of Life in Patients With Unicompartmental Arthrosis After High Tibial Osteotomy With the Position HTO(R) System
Brief Title: Position HTO Multicenter NIS
Acronym: Position HTO
Status: Completed | Type: Observational
Sponsor: Aesculap AG (Industry)
Responsible Party: Viktor Breul, Aesculap AG
Other Study IDs: AAG-O-H-0702
Record Dates: First submitted 2009-04-27; First posted 2009-04-28 (Estimated); Last update posted 2011-07-22 (Estimated); Status verified 2011-07

CONDITIONS: Medial Monocompartmental Osteoarthritis of the Knee
Keywords: HTO, high tibial osteotomy, open wedge, medial arthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- A: HTO cohort
  Interventions: Device: Position HTO system

INTERVENTIONS:
Device: Position HTO system — open wedge high tibial osteotomy

SUMMARY:
Evaluation of the Position HTO system in patients with unicompartmental medial arthrosis after open wedge high tibial osteotomy

ELIGIBILITY:
Inclusion: Varus deformity between 0 - 20°, Isolated medial arthrosis ≥ level 2 (K&L) OR a congenital deformity OR chondromalacia ≥ level 2 (ICRS), Lateral cartilaginous tissue damage ≤ level 1(K&L), Intact lateral meniscus, Age ≥ 18 years, Range of Motion at least 0° - 0° - 130°, Patella/ sliding plane without signifikant signs of arthrosis, Stable joint OR possibility of intraoperative balancing of the tendon tension;

Exclusion: Clinically relevant disorders of bone metabolism, Aktive infection, Adipositas (BMI ≥ 35), Rheumatoid arthritis, Osteomyelitis in the tibia, No availibility for follow-up examinations

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adult patients
Sampling Method: Probability Sample
Enrollment: 221 (Actual)
Dates: Start 2007-07; Primary Completion 2009-08 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Patient health status improvement assessed by IKDC 2000 subjective knee score | 1 year after HTO

SECONDARY OUTCOMES:
Improvement of further scores: Tegner Activity Score, Lysholm-Gillquist Score, Cincinnati-Sportsmedicine and Orthopaedic Center-Score, IKDC 2000 objective knee score, Hospital for Special Surgery Score (HSS) | 1 year after HTO

CONTACTS AND LOCATIONS:
Overall Officials: Jürgen Fritz, Dr., Principal Investigator — Winghofer Medicum
Locations (5):
- Germany (5):
  - Orthopädie Harthausen, Bad Aibling
  - Caritas-Krankenhaus Bad Mergentheim, Bad Mergentheim
  - Universitätsklinikum Regensburg, Regensburg
  - Winghofer Medicum, Rottenburg
  - BGU Tübingen, Tübingen